CLINICAL TRIAL: NCT04583618
Title: Safety and Immunogenicity of a Pneumococcal Conjugate Vaccine in Healthy Adults Aged 50 to 84 Years
Brief Title: Study of a Pneumococcal Conjugate Vaccine in Adults Aged 50 to 84 Years.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK00009; U1111-1238-9824 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Immunization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- SP0202-IIb (Experimental): One dose at Day 1
  Interventions: Biological: Pneumococcal Conjugate Vaccine - formulation 1-SP0202-IIb
- SP0202-VI (Experimental): One dose at Day 1
  Interventions: Biological: Pneumococcal Conjugate Vaccine - formulation 2-SP0202-VI
- SP0202-VII (Experimental): One dose at Day 1
  Interventions: Biological: Pneumococcal Conjugate Vaccine - formulation 3-SP0202-VII
- Prevnar 13 (Active Comparator): One dose at Day 1
  Interventions: Biological: Pneumococcal 13 - valent conjugate vaccine-Prevnar 13
- Pneumovax 23 (Active Comparator): One dose at Day 1
  Interventions: Biological: Pneumococcal Vaccine Polyvalent-Pneumovax 23

INTERVENTIONS:
Biological: Pneumococcal Conjugate Vaccine - formulation 1-SP0202-IIb — Pharmaceutical form:Suspension for injection Route of administration: intramuscular
  Arms: SP0202-IIb
Biological: Pneumococcal Conjugate Vaccine - formulation 2-SP0202-VI — Pharmaceutical form:Suspension for injection Route of administration: intramuscular
  Arms: SP0202-VI
Biological: Pneumococcal Conjugate Vaccine - formulation 3-SP0202-VII — Pharmaceutical form:Suspension for injection Route of administration: intramuscular
  Arms: SP0202-VII
Biological: Pneumococcal 13 - valent conjugate vaccine-Prevnar 13 — Pharmaceutical form:Suspension for injection Route of administration: intramuscular
  Arms: Prevnar 13
Biological: Pneumococcal Vaccine Polyvalent-Pneumovax 23 — Pharmaceutical form:Solution for injection Route of administration: intramuscular
  Arms: Pneumovax 23

SUMMARY:
Primary Objectives:

* Assessed the immune response of the 3 SP0202 formulations, Prevnar 13 and Pneumovax 23 30 days after the administration of the single dose vaccination
* Assessed the safety profile of the 3 SP0202 formulations, Prevnar 13 and Pneumovax 23

DETAILED DESCRIPTION:
The duration of each participant's participation was approximately 6 months.

ELIGIBILITY:
Inclusion criteria :

- Aged 50 to 84 years on the day of inclusion .

Exclusion criteria:

* Participant was pregnant, or lactating, or of childbearing potential and was not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, the female must have been post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of the study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device or medical procedure.
* Received any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine from enrollment through the last blood sampling Visit, except for influenza vaccination, which may be received at least 2 weeks before study vaccine. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against S. pneumoniae with either a pneumococcal conjugated vaccine (PCV) or a pneumococcal polysaccharide vaccine (PPSV).
* Received immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of S. pneumoniae infection or disease, confirmed either serologically, or microbiologically.
* History of Guillain-Barré syndrome occurring within 6 weeks after a prior dose of a TTxd-containing vaccine.
* Experienced an Arthus-type hypersensitivity reaction following a prior dose of a TTxd-containing vaccine < 10 years ago.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances .
* Verbal report of thrombocytopenia contraindicating IM vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination in the Investigator's opinion.
* At risk of invasive pneumococcal disease (eg, participants with functional or anatomic asplenia, participants with severe asthma, participants travelling to countries with high endemicity).
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Any condition that in the opinion of the Investigator could interfere with the evaluation of the vaccine (eg, under investigation or monitoring for possible coronavirus disease 2019 [COVID-19]).
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4 F). A prospective participant should not be included in the study until the condition has resolved or until 3 days after the febrile event has subsided.
* Received oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- United States (17):
  - Emmaus Research Center, Inc Site Number : 8400014, Anaheim, California
  - Peninsula Research Associates Site Number : 8400012, Rolling Hills Estates, California
  - Paradigm Clinical Research Center Wheat Ridge Site Number : 8400002, Wheat Ridge, Colorado
  - Jacksonville Center for Clinical Research Site Number : 8400016, Jacksonville, Florida
  - Suncoast Research Associates, LLC Site Number : 8400017, Miami, Florida
  - Advanced Clinical Research - Magic View Site Number : 8400003, Meridian, Idaho
  - Velocity Clinical Research Valparaiso Site Number : 8400001, Valparaiso, Indiana
  - Velocity Clinical Research Site Number : 8400005, Metairie, Louisiana
  - Be Well Clinical Studies Site Number : 8400018, Lincoln, Nebraska
  - WR-CRCN, LLC Site Number : 8400013, Las Vegas, Nevada
  - Biotrial Inc Site Number : 8400006, Newark, New Jersey
  - Plains Clinical Research Center, LLC Site Number : 8400011, Fargo, North Dakota
  - Aventiv Research Columbus Site Number : 8400007, Columbus, Ohio
  - Velocity Clinical Research, Medford Site Number : 8400010, Medford, Oregon
  - Preferred Primary Care Physicians Site Number : 8400009, Pittsburgh, Pennsylvania
  - Coastal Carolina Research Center - N Charleston Site Number : 8400004, North Charleston, South Carolina
  - JBR Clinical Research Site Number : 8400008, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PSK00009 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25337&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 investigational sites in United States between 08 Oct 2020 to 20 Jan 2022.
Pre-assignment Details: A total of 750 participants were enrolled in this study.
Groups:
- Group 1: SP0202-IIb: Healthy participants aged 50 to 84 years who were naïve to previous pneumococcal vaccination received a single intramuscular (IM) injection of SP0202-IIb formulation at Day 1.
- Group 2: SP0202-VI: Healthy participants aged 50 to 84 years who were naïve to previous pneumococcal vaccination received a single IM injection of SP0202-VI formulation at Day 1.
- Group 3: SP0202-VII: Healthy participants aged 50 to 84 years who were naïve to previous pneumococcal vaccination received a single IM injection of SP0202-VII formulation at Day 1.
- Group 4: Prevnar 13: Healthy participants aged 50 to 84 years who were naïve to previous pneumococcal vaccination received a single IM injection of Prevnar 13 at Day 1.
- Group 5: Pneumovax 23: Healthy participants aged 50 to 84 years who were naïve to previous pneumococcal vaccination received a single IM injection of Pneumovax 23 at Day 1.
Period: Overall Study
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Started | 151 | 151 | 149 | 149 | 150
Safety Analysis Set (SafAS) Population | 151 | 151 | 148 | 149 | 150
Completed | 148 | 148 | 141 | 147 | 148
Not Completed | 3 | 3 | 8 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants with data in the case report form (CRF).
Groups:
- Group 1: SP0202-IIb: Healthy participants aged 50 to 84 years who were naïve to previous pneumococcal vaccination received a single IM injection of SP0202-IIb formulation at Day 1.
- Total: Total of all reporting groups
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23 | Total
Number analyzed (Participants) | 151 | 151 | 149 | 149 | 150 | 750
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (6.9) | 63.1 (6.6) | 62.9 (6.5) | 63.4 (6.8) | 63.1 (7.2) | 63.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 84 | 78 | 86 | 93 | 417
  Male | 75 | 67 | 71 | 63 | 57 | 333
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 1 | 0 | 4
  Black or African American | 19 | 17 | 24 | 10 | 13 | 83
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1 | 0 | 2
  White | 120 | 123 | 113 | 127 | 121 | 604
  Asian | 10 | 9 | 9 | 10 | 11 | 49
  Multiple | 1 | 0 | 0 | 0 | 1 | 2
  Not reported | 0 | 1 | 1 | 0 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Pneumococcal Serotypes Using Serotype-Specific MOPA
Description: The GMs for serotype specific OPA titers were measured using MOPA which was used to evaluate the opsonophagocytic index (50% killing) of pneumococcal anti-capsular polysaccharide antibodies in human serum samples following vaccination. Titers were expressed in terms of 1/dilution.
Time Frame: Post-vaccination at Day 31
Population: PPAS was subset of the FAS. FAS included subset of randomized participants who received at least 1 dose of the study vaccine and had a valid post-vaccination blood sample result (serotype specific IgG concentration or serotype specific OPA titer for at least one serotype). Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 135 | 143 | 134 | 139 | 136
Titer
  Serotype 1: number analyzed (Participants) | 135 | 142 | 134 | 137 | 135
  Serotype 1 | 128 [92.5 to 177] | 127 [90.3 to 178] | 158 [113 to 220] | 254 [183 to 353] | 289 [213 to 392]
  Serotype 3: number analyzed (Participants) | 135 | 142 | 134 | 138 | 135
  Serotype 3 | 136 [109 to 170] | 217 [176 to 269] | 263 [214 to 323] | 157 [126 to 196] | 177 [142 to 221]
  Serotype 4 | 1494 [1175 to 1900] | 1306 [1029 to 1658] | 2134 [1675 to 2719] | 2941 [2360 to 3664] | 1873 [1415 to 2480]
  Serotype 5 | 241 [166 to 349] | 230 [160 to 330] | 201 [143 to 281] | 536 [378 to 760] | 377 [272 to 523]
  Serotype 6A: number analyzed (Participants) | 135 | 142 | 133 | 135 | 134
  Serotype 6A | 2931 [2143 to 4010] | 3074 [2389 to 3957] | 2672 [1923 to 3714] | 3350 [2418 to 4641] | 443 [288 to 681]
  Serotype 6B: number analyzed (Participants) | 134 | 143 | 134 | 139 | 136
  Serotype 6B | 3699 [2857 to 4788] | 3582 [2763 to 4645] | 3479 [2595 to 4664] | 5122 [3916 to 6699] | 2153 [1561 to 2969]
  Serotype 7F | 3487 [2811 to 4326] | 2841 [2262 to 3568] | 2403 [1878 to 3074] | 4253 [3309 to 5466] | 2250 [1721 to 2943]
  Serotype 9V: number analyzed (Participants) | 135 | 142 | 134 | 139 | 136
  Serotype 9V | 826 [607 to 1123] | 828 [614 to 1117] | 986 [700 to 1388] | 1641 [1274 to 2114] | 1159 [863 to 1556]
  Serotype 14 | 3756 [2995 to 4709] | 4407 [3385 to 5737] | 3244 [2421 to 4349] | 3675 [2904 to 4650] | 3999 [3099 to 5161]
  Serotype 18C | 905 [676 to 1210] | 802 [590 to 1090] | 1025 [756 to 1390] | 1929 [1460 to 2548] | 1177 [875 to 1585]
  Serotype 19A | 2067 [1719 to 2485] | 3395 [2796 to 4123] | 3462 [2771 to 4324] | 4417 [3537 to 5515] | 2261 [1841 to 2776]
  Serotype 19F: number analyzed (Participants) | 134 | 143 | 134 | 139 | 136
  Serotype 19F | 897 [702 to 1145] | 1773 [1406 to 2236] | 1678 [1336 to 2108] | 1525 [1165 to 1997] | 983 [742 to 1303]
  Serotype 23F: number analyzed (Participants) | 135 | 143 | 134 | 138 | 135
  Serotype 23F | 1999 [1478 to 2704] | 1576 [1153 to 2153] | 1701 [1284 to 2255] | 1792 [1311 to 2450] | 488 [319 to 747]
  Serotype 8 | 1363 [1110 to 1674] | 1377 [1129 to 1680] | 1486 [1207 to 1829] | 74.8 [52.3 to 107] | 2039 [1664 to 2499]
  Serotype 9N: number analyzed (Participants) | 135 | 142 | 133 | 137 | 136
  Serotype 9N | 3656 [2988 to 4474] | 3858 [3145 to 4733] | 4207 [3430 to 5160] | 1082 [806 to 1453] | 6096 [4837 to 7682]
  Serotype 10A: number analyzed (Participants) | 135 | 143 | 133 | 135 | 133
  Serotype 10A | 3501 [2689 to 4557] | 2856 [2190 to 3724] | 2811 [2047 to 3860] | 104 [64.3 to 167] | 3011 [2060 to 4399]
  Serotype 11A: number analyzed (Participants) | 134 | 142 | 134 | 137 | 136
  Serotype 11A | 475 [354 to 637] | 438 [324 to 594] | 318 [226 to 448] | 18.3 [13.0 to 25.6] | 390 [285 to 534]
  Serotype 12F: number analyzed (Participants) | 135 | 143 | 134 | 136 | 135
  Serotype 12F | 3492 [2587 to 4714] | 3917 [3116 to 4925] | 3117 [2311 to 4203] | 8.31 [6.19 to 11.2] | 1345 [914 to 1980]
  Serotype 15B: number analyzed (Participants) | 134 | 140 | 130 | 136 | 132
  Serotype 15B | 4930 [3641 to 6677] | 4823 [3588 to 6484] | 3613 [2541 to 5138] | 160 [112 to 230] | 3346 [2409 to 4648]
  Serotype 22F: number analyzed (Participants) | 135 | 140 | 132 | 134 | 133
  Serotype 22F | 5253 [4147 to 6653] | 4639 [3587 to 6001] | 4858 [3683 to 6406] | 62.5 [42.4 to 92.1] | 1906 [1456 to 2495]
  Serotype 33F: number analyzed (Participants) | 135 | 143 | 134 | 138 | 136
  Serotype 33F | 7313 [5890 to 9078] | 8324 [6488 to 10680] | 7641 [6205 to 9410] | 1201 [898 to 1605] | 15082 [11551 to 19692]

2. Primary Outcome: Geometric Mean Titers Ratio of Pneumococcal Serotypes Using Serotype-Specific MOPA
Description: The GMs for serotype specific OPA titers were measured using MOPA which was used to evaluate the opsonophagocytic index (50% killing) of pneumococcal anti-capsular polysaccharide antibodies in human serum samples following vaccination. Ratio was calculated as post-vaccination titer at Day 31 to pre-vaccination titer at Day 1.
Time Frame: Pre-vaccination at Baseline (Day 1) and Post-vaccination at Day 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 135 | 143 | 134 | 138 | 136
Ratio
  Serotype 1: number analyzed (Participants) | 135 | 142 | 134 | 136 | 134
  Serotype 1 | 8.40 [6.28 to 11.2] | 10.5 [7.95 to 14.0] | 9.79 [7.15 to 13.4] | 21.3 [15.6 to 29.0] | 19.1 [14.4 to 25.3]
  Serotype 3: number analyzed (Participants) | 135 | 142 | 131 | 136 | 135
  Serotype 3 | 7.06 [5.55 to 8.99] | 12.9 [10.1 to 16.4] | 13.7 [10.7 to 17.4] | 8.52 [6.71 to 10.8] | 9.52 [7.56 to 12.0]
  Serotype 4: number analyzed (Participants) | 134 | 142 | 134 | 136 | 135
  Serotype 4 | 20.7 [14.7 to 29.3] | 28.8 [20.6 to 40.3] | 33.0 [22.2 to 49.2] | 58.9 [41.2 to 84.1] | 25.7 [18.2 to 36.4]
  Serotype 5 | 15.2 [11.0 to 21.0] | 19.5 [14.3 to 26.7] | 12.2 [9.10 to 16.4] | 37.4 [26.9 to 52.1] | 24.2 [18.2 to 32.2]
  Serotype 6A: number analyzed (Participants) | 135 | 141 | 133 | 134 | 132
  Serotype 6A | 60.8 [42.8 to 86.5] | 69.4 [48.3 to 99.8] | 59.2 [40.9 to 85.8] | 79.1 [54.4 to 115] | 9.18 [6.34 to 13.3]
  Serotype 6B: number analyzed (Participants) | 134 | 140 | 133 | 136 | 133
  Serotype 6B | 29.1 [20.6 to 41.2] | 25.7 [18.1 to 36.6] | 29.2 [19.5 to 43.6] | 49.3 [34.8 to 69.7] | 16.6 [11.5 to 23.8]
  Serotype 7F: number analyzed (Participants) | 132 | 141 | 132 | 138 | 134
  Serotype 7F | 50.8 [32.8 to 78.9] | 49.0 [32.5 to 73.7] | 24.0 [14.9 to 38.7] | 79.1 [51.6 to 121] | 31.0 [21.0 to 45.8]
  Serotype 9V: number analyzed (Participants) | 133 | 141 | 134 | 138 | 135
  Serotype 9V | 9.50 [7.01 to 12.9] | 9.90 [7.20 to 13.6] | 12.7 [8.90 to 18.0] | 17.2 [12.2 to 24.1] | 10.6 [7.78 to 14.4]
  Serotype 14: number analyzed (Participants) | 133 | 141 | 134 | 138 | 136
  Serotype 14 | 7.44 [5.25 to 10.5] | 14.3 [9.69 to 21.0] | 8.44 [5.68 to 12.5] | 10.1 [7.03 to 14.6] | 9.05 [6.46 to 12.7]
  Serotype 18C: number analyzed (Participants) | 135 | 142 | 134 | 138 | 136
  Serotype 18C | 17.0 [12.4 to 23.3] | 20.6 [15.0 to 28.2] | 18.9 [13.3 to 27.0] | 43.1 [31.1 to 59.8] | 22.1 [16.3 to 30.0]
  Serotype 19A | 7.36 [5.77 to 9.38] | 13.1 [10.3 to 16.8] | 11.5 [8.66 to 15.3] | 15.5 [11.4 to 21.0] | 7.88 [6.26 to 9.91]
  Serotype 19F: number analyzed (Participants) | 134 | 142 | 134 | 138 | 136
  Serotype 19F | 13.1 [9.45 to 18.2] | 30.7 [21.9 to 43.0] | 20.8 [15.0 to 29.0] | 26.6 [19.0 to 37.1] | 17.2 [12.5 to 23.7]
  Serotype 23F: number analyzed (Participants) | 134 | 141 | 133 | 135 | 133
  Serotype 23F | 45.2 [31.0 to 65.9] | 43.0 [29.0 to 63.8] | 43.9 [29.6 to 65.1] | 45.5 [32.2 to 64.4] | 11.6 [7.99 to 16.8]
  Serotype 8: number analyzed (Participants) | 134 | 140 | 133 | 138 | 135
  Serotype 8 | 18.6 [13.5 to 25.6] | 24.1 [17.7 to 32.8] | 24.0 [16.3 to 35.3] | 1.37 [1.14 to 1.65] | 37.6 [27.8 to 50.8]
  Serotype 9N: number analyzed (Participants) | 132 | 136 | 127 | 131 | 133
  Serotype 9N | 8.90 [6.29 to 12.6] | 12.8 [8.90 to 18.4] | 11.5 [7.88 to 16.8] | 2.84 [2.12 to 3.79] | 14.6 [10.7 to 20.0]
  Serotype 10A: number analyzed (Participants) | 135 | 139 | 131 | 134 | 130
  Serotype 10A | 24.2 [16.3 to 35.8] | 24.7 [16.5 to 36.9] | 20.8 [13.4 to 32.3] | 1.05 [0.932 to 1.19] | 22.9 [16.1 to 32.7]
  Serotype 11A: number analyzed (Participants) | 132 | 138 | 130 | 132 | 136
  Serotype 11A | 14.8 [10.4 to 21.0] | 15.9 [11.1 to 22.6] | 9.28 [6.46 to 13.3] | 0.964 [0.786 to 1.18] | 13.7 [9.64 to 19.5]
  Serotype 12F: number analyzed (Participants) | 132 | 140 | 133 | 133 | 134
  Serotype 12F | 240 [163 to 354] | 252 [181 to 353] | 167 [106 to 263] | 0.975 [0.870 to 1.09] | 102 [67.7 to 153]
  Serotype 15B: number analyzed (Participants) | 133 | 133 | 127 | 130 | 128
  Serotype 15B | 30.1 [20.8 to 43.6] | 34.3 [23.3 to 50.5] | 20.7 [14.1 to 30.4] | 1.21 [0.997 to 1.47] | 22.8 [16.1 to 32.1]
  Serotype 22F: number analyzed (Participants) | 127 | 135 | 129 | 130 | 129
  Serotype 22F | 39.0 [27.2 to 56.1] | 41.4 [28.5 to 60.3] | 38.5 [25.4 to 58.3] | 0.878 [0.679 to 1.14] | 21.0 [15.1 to 29.1]
  Serotype 33F: number analyzed (Participants) | 133 | 139 | 132 | 137 | 134
  Serotype 33F | 4.21 [3.27 to 5.41] | 6.27 [4.72 to 8.32] | 4.36 [3.45 to 5.52] | 0.931 [0.871 to 0.995] | 10.4 [7.76 to 13.9]

3. Primary Outcome: Geometric Mean Concentrations (GMCs) of Pneumococcal Serotypes Using Serotype-Specific IgG ECL
Description: The GMCs for serotype specific pneumococcal IgG antibodies were measured using ECL, a multiplexed serological assay which allowed for the simultaneous quantification of human IgG against pneumococcal polysaccharide antigens.
Time Frame: Post-vaccination at Day 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 137 | 144 | 134 | 139 | 141
mcg/mL
  Serotype 1 | 2.98 [2.29 to 3.88] | 3.28 [2.59 to 4.17] | 4.17 [3.29 to 5.28] | 5.93 [4.49 to 7.85] | 7.43 [5.75 to 9.60]
  Serotype 3: number analyzed (Participants) | 137 | 143 | 133 | 139 | 141
  Serotype 3 | 0.746 [0.616 to 0.903] | 0.977 [0.818 to 1.17] | 1.22 [1.01 to 1.49] | 0.899 [0.738 to 1.10] | 0.858 [0.717 to 1.03]
  Serotype 4 | 1.97 [1.60 to 2.43] | 1.63 [1.32 to 2.00] | 2.27 [1.81 to 2.84] | 3.28 [2.61 to 4.12] | 1.72 [1.38 to 2.13]
  Serotype 5: number analyzed (Participants) | 136 | 144 | 134 | 139 | 141
  Serotype 5 | 2.35 [1.78 to 3.10] | 2.16 [1.62 to 2.87] | 2.16 [1.68 to 2.78] | 4.34 [3.20 to 5.90] | 3.98 [3.09 to 5.12]
  Serotype 6A: number analyzed (Participants) | 137 | 144 | 134 | 138 | 141
  Serotype 6A | 6.04 [4.45 to 8.22] | 5.00 [3.83 to 6.54] | 4.83 [3.57 to 6.54] | 7.89 [5.90 to 10.5] | 1.53 [1.16 to 2.02]
  Serotype 6B | 5.73 [4.17 to 7.89] | 3.62 [2.66 to 4.93] | 4.37 [3.22 to 5.95] | 6.45 [4.92 to 8.45] | 2.47 [1.86 to 3.28]
  Serotype 7F | 6.56 [5.23 to 8.22] | 5.56 [4.58 to 6.75] | 5.35 [4.30 to 6.65] | 10.1 [8.01 to 12.6] | 4.23 [3.34 to 5.35]
  Serotype 9V | 2.91 [2.29 to 3.72] | 3.17 [2.52 to 4.00] | 4.31 [3.43 to 5.41] | 5.30 [4.20 to 6.68] | 3.48 [2.75 to 4.41]
  Serotype 14: number analyzed (Participants) | 137 | 143 | 134 | 138 | 140
  Serotype 14 | 12.4 [9.88 to 15.7] | 10.5 [8.21 to 13.6] | 9.52 [7.34 to 12.3] | 10.5 [8.22 to 13.4] | 14.6 [11.2 to 19.0]
  Serotype 18C | 5.50 [4.44 to 6.82] | 5.39 [4.39 to 6.62] | 5.41 [4.44 to 6.59] | 10.3 [8.15 to 13.1] | 5.44 [4.34 to 6.81]
  Serotype 19A | 7.41 [6.03 to 9.10] | 11.7 [9.16 to 15.1] | 10.9 [8.41 to 14.2] | 18.3 [14.4 to 23.2] | 7.59 [6.05 to 9.52]
  Serotype 19F: number analyzed (Participants) | 137 | 144 | 134 | 138 | 141
  Serotype 19F | 3.77 [2.92 to 4.87] | 8.35 [6.22 to 11.2] | 7.03 [5.30 to 9.33] | 9.38 [7.16 to 12.3] | 4.47 [3.40 to 5.88]
  Serotype 23F | 7.35 [5.56 to 9.72] | 5.52 [4.26 to 7.13] | 6.59 [5.05 to 8.61] | 6.99 [5.33 to 9.17] | 3.02 [2.31 to 3.96]
  Serotype 8: number analyzed (Participants) | 137 | 144 | 134 | 136 | 141
  Serotype 8 | 7.14 [5.75 to 8.87] | 6.25 [5.09 to 7.68] | 6.23 [4.98 to 7.80] | 0.935 [0.703 to 1.24] | 9.84 [8.14 to 11.9]
  Serotype 9N | 5.26 [4.06 to 6.81] | 4.50 [3.55 to 5.71] | 6.54 [5.09 to 8.40] | 1.60 [1.20 to 2.12] | 6.41 [5.10 to 8.06]
  Serotype 10A: number analyzed (Participants) | 137 | 144 | 134 | 138 | 140
  Serotype 10A | 7.16 [5.37 to 9.55] | 9.48 [7.10 to 12.6] | 7.37 [5.39 to 10.1] | 1.06 [0.840 to 1.35] | 9.11 [6.83 to 12.1]
  Serotype 11A | 4.85 [3.99 to 5.89] | 4.91 [4.08 to 5.89] | 4.27 [3.51 to 5.20] | 0.884 [0.745 to 1.05] | 3.88 [3.19 to 4.72]
  Serotype 12F | 2.18 [1.58 to 3.02] | 2.09 [1.55 to 2.83] | 1.90 [1.41 to 2.55] | 0.190 [0.158 to 0.228] | 1.03 [0.780 to 1.36]
  Serotype 15B: number analyzed (Participants) | 137 | 144 | 133 | 139 | 141
  Serotype 15B | 13.4 [10.5 to 17.2] | 16.3 [12.8 to 20.8] | 14.8 [11.7 to 18.8] | 1.84 [1.42 to 2.39] | 13.6 [10.8 to 17.2]
  Serotype 22F | 3.57 [2.88 to 4.44] | 4.02 [3.20 to 5.05] | 3.78 [3.03 to 4.71] | 0.350 [0.283 to 0.433] | 2.41 [1.93 to 3.00]
  Serotype 33F | 7.98 [6.19 to 10.3] | 9.15 [7.42 to 11.3] | 7.75 [6.18 to 9.72] | 1.50 [1.21 to 1.85] | 16.4 [12.8 to 21.1]

4. Primary Outcome: Geometric Mean Concentrations Ratio of Pneumococcal Serotypes Using Serotype-Specific IgG ECL
Description: The GMCs for serotype specific pneumococcal IgG antibodies were measured using ECL, a multiplexed serological assay which allowed for the simultaneous quantification of human IgG against pneumococcal polysaccharide antigens. Ratio was calculated as post-vaccination titer at Day 31 to pre-vaccination titer at Day 1.
Time Frame: Pre-vaccination at Baseline (Day 1) and Post-vaccination at Day 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 137 | 144 | 134 | 139 | 141
Ratio
  Serotype 1 | 5.39 [4.33 to 6.70] | 6.47 [5.27 to 7.95] | 6.41 [5.11 to 8.03] | 11.6 [9.21 to 14.6] | 11.5 [9.09 to 14.5]
  Serotype 3: number analyzed (Participants) | 137 | 143 | 132 | 139 | 141
  Serotype 3 | 2.99 [2.49 to 3.61] | 4.02 [3.40 to 4.76] | 4.93 [4.07 to 5.97] | 3.86 [3.21 to 4.65] | 3.52 [3.01 to 4.12]
  Serotype 4 | 6.52 [5.32 to 7.98] | 5.91 [4.93 to 7.07] | 7.33 [5.90 to 9.10] | 10.8 [8.71 to 13.3] | 5.47 [4.57 to 6.55]
  Serotype 5: number analyzed (Participants) | 136 | 144 | 134 | 139 | 141
  Serotype 5 | 5.43 [4.32 to 6.82] | 5.81 [4.67 to 7.22] | 4.60 [3.75 to 5.66] | 10.6 [8.15 to 13.7] | 8.93 [7.15 to 11.1]
  Serotype 6A: number analyzed (Participants) | 137 | 144 | 134 | 138 | 141
  Serotype 6A | 13.8 [10.5 to 18.2] | 12.2 [9.79 to 15.3] | 12.6 [9.76 to 16.4] | 19.3 [14.9 to 24.9] | 3.30 [2.75 to 3.96]
  Serotype 6B | 12.2 [9.31 to 16.0] | 9.63 [7.59 to 12.2] | 10.7 [8.10 to 14.0] | 16.2 [12.8 to 20.5] | 5.51 [4.51 to 6.74]
  Serotype 7F: number analyzed (Participants) | 137 | 143 | 134 | 139 | 141
  Serotype 7F | 10.6 [8.37 to 13.4] | 9.67 [7.86 to 11.9] | 7.93 [6.30 to 9.99] | 16.3 [12.8 to 20.7] | 6.80 [5.67 to 8.16]
  Serotype 9V | 5.65 [4.59 to 6.95] | 6.29 [5.09 to 7.76] | 7.87 [6.28 to 9.86] | 9.12 [7.53 to 11.0] | 6.30 [5.17 to 7.68]
  Serotype 14: number analyzed (Participants) | 137 | 142 | 134 | 138 | 139
  Serotype 14 | 4.91 [3.93 to 6.13] | 6.44 [5.06 to 8.19] | 4.62 [3.59 to 5.95] | 5.96 [4.68 to 7.58] | 7.35 [5.85 to 9.23]
  Serotype 18C | 6.52 [5.26 to 8.08] | 7.18 [5.86 to 8.79] | 6.21 [5.09 to 7.58] | 12.1 [9.52 to 15.3] | 6.91 [5.74 to 8.31]
  Serotype 19A | 4.74 [3.89 to 5.78] | 8.76 [7.14 to 10.7] | 7.86 [6.28 to 9.84] | 12.3 [9.79 to 15.4] | 5.74 [4.72 to 6.98]
  Serotype 19F: number analyzed (Participants) | 137 | 144 | 133 | 138 | 141
  Serotype 19F | 4.97 [4.02 to 6.15] | 11.2 [8.82 to 14.3] | 9.65 [7.53 to 12.4] | 11.2 [8.77 to 14.2] | 6.18 [5.07 to 7.53]
  Serotype 23F | 13.2 [10.2 to 17.2] | 11.0 [8.75 to 13.9] | 11.9 [9.21 to 15.3] | 13.0 [10.3 to 16.4] | 5.70 [4.57 to 7.12]
  Serotype 8: number analyzed (Participants) | 137 | 144 | 134 | 136 | 141
  Serotype 8 | 7.97 [6.41 to 9.92] | 8.44 [6.88 to 10.3] | 8.20 [6.54 to 10.3] | 1.26 [1.11 to 1.42] | 13.9 [11.5 to 16.8]
  Serotype 9N: number analyzed (Participants) | 137 | 144 | 134 | 139 | 140
  Serotype 9N | 6.52 [5.22 to 8.14] | 8.39 [6.67 to 10.5] | 9.99 [7.87 to 12.7] | 2.81 [2.36 to 3.35] | 11.3 [9.20 to 13.8]
  Serotype 10A: number analyzed (Participants) | 137 | 144 | 134 | 138 | 140
  Serotype 10A | 8.45 [6.74 to 10.6] | 10.0 [8.01 to 12.6] | 7.55 [5.83 to 9.78] | 1.15 [1.07 to 1.22] | 9.84 [7.98 to 12.1]
  Serotype 11A | 5.57 [4.56 to 6.82] | 6.13 [5.08 to 7.38] | 5.36 [4.36 to 6.61] | 1.18 [1.10 to 1.27] | 5.54 [4.65 to 6.60]
  Serotype 12F | 8.70 [6.66 to 11.4] | 9.47 [7.29 to 12.3] | 8.05 [6.20 to 10.5] | 1.08 [1.02 to 1.14] | 5.07 [4.01 to 6.40]
  Serotype 15B: number analyzed (Participants) | 137 | 144 | 133 | 139 | 141
  Serotype 15B | 7.77 [6.28 to 9.63] | 11.6 [9.13 to 14.7] | 8.74 [6.99 to 10.9] | 1.35 [1.19 to 1.52] | 9.87 [7.95 to 12.2]
  Serotype 22F | 9.21 [7.38 to 11.5] | 10.0 [8.09 to 12.5] | 8.99 [7.32 to 11.0] | 1.09 [1.02 to 1.17] | 7.30 [5.95 to 8.95]
  Serotype 33F | 4.54 [3.68 to 5.60] | 5.59 [4.58 to 6.81] | 4.43 [3.60 to 5.45] | 1.03 [0.981 to 1.08] | 9.43 [7.64 to 11.6]

5. Primary Outcome: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the CRF in terms of diagnosis and/or onset window post-vaccination. Systemic AEs were all AEs that were not injection or administration site reactions.
Time Frame: Within 30 minutes post-vaccination
Population: Safety analysis set (SafAS) included participants who had received the study vaccine. All participants had their safety analyzed according to the vaccine they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 151 | 151 | 148 | 149 | 150
Participants | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. An injection site reaction was an AR at and around the injection site. Solicited injection site reactions included injection site pain, injection site erythema and injection site swelling.
Time Frame: Up to 7 Days post-vaccination (Day 8)
Population: SafAS included participants who had received the study vaccine. All participants had their safety analyzed according to the vaccine they actually received. Only those participants with data collected for each category at each specified timepoint are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 149 | 149 | 141 | 146 | 150
Participants
  Injection site pain | 106 | 113 | 107 | 85 | 74
  Injection site erythema | 17 | 25 | 19 | 3 | 9
  Injection site swelling | 14 | 19 | 14 | 4 | 6

7. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. Solicited systemic reactions included fever, headache, malaise, myalgia, arthralgia and shivering.
Time Frame: Up to 7 Days post-vaccination (Day 8)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 149 | 149 | 141 | 146 | 150
Participants
  Fever: number analyzed (Participants) | 146 | 145 | 139 | 145 | 150
  Fever | 3 | 2 | 5 | 3 | 4
  Headache | 43 | 47 | 38 | 35 | 41
  Malaise | 36 | 43 | 30 | 28 | 32
  Myalgia | 57 | 71 | 56 | 49 | 65
  Arthralgia | 23 | 30 | 18 | 17 | 29
  Shivering | 20 | 27 | 18 | 7 | 13

8. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the CRF in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Within 30 days post-vaccination
Population: SafAS included participants who had received the study vaccine. All participants had their safety analyzed according to the vaccine they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 151 | 151 | 148 | 149 | 150
Participants | 21 | 34 | 19 | 18 | 20

9. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Event of Special Interest (AESIs)
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI was defined as one of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor could be appropriate. AESI included analyphylaxis.
Time Frame: From the study vaccine administration (Day 1) until the end of 6-Month follow-up, 181 days
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
Number analyzed (Participants) | 151 | 151 | 148 | 149 | 150
Participants
  SAEs | 3 | 7 | 3 | 2 | 2
  AESIs | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs, SAEs and all-cause mortality (deaths) were collected from the study vaccine administration (Day 1) until the end of 6-Month follow-up, 181 days.
Description: Analysis was performed on SafAS.
Arm/Group | Group 1: SP0202-IIb | Group 2: SP0202-VI | Group 3: SP0202-VII | Group 4: Prevnar 13 | Group 5: Pneumovax 23
All-Cause Mortality (participants affected / at risk) | 0/151 | 1/151 | 1/148 | 0/149 | 0/150
Serious Adverse Events (participants affected / at risk) | 3/151 | 7/151 | 3/148 | 2/149 | 2/150
Other Adverse Events (participants affected / at risk) | 113/151 | 122/151 | 112/148 | 102/149 | 93/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: SP0202-IIb (N=151) | Group 2: SP0202-VI (N=151) | Group 3: SP0202-VII (N=148) | Group 4: Prevnar 13 (N=149) | Group 5: Pneumovax 23 (N=150)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: SP0202-IIb (N=151) | Group 2: SP0202-VI (N=151) | Group 3: SP0202-VII (N=148) | Group 4: Prevnar 13 (N=149) | Group 5: Pneumovax 23 (N=150)
Chills (General disorders) | 20 (20) | 27 (27) | 18 (18) | 7 (7) | 13 (13)
Injection Site Erythema (General disorders) | 17 (18) | 25 (25) | 20 (20) | 4 (4) | 9 (10)
Injection Site Pain (General disorders) | 106 (106) | 113 (113) | 107 (107) | 85 (85) | 74 (74)
Injection Site Swelling (General disorders) | 14 (15) | 19 (19) | 14 (14) | 4 (4) | 6 (6)
Malaise (General disorders) | 36 (36) | 43 (43) | 30 (30) | 28 (28) | 32 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (23) | 30 (30) | 18 (18) | 17 (17) | 31 (31)
Myalgia (Musculoskeletal and connective tissue disorders) | 57 (58) | 72 (72) | 56 (56) | 49 (50) | 65 (65)
Headache (Nervous system disorders) | 43 (43) | 48 (51) | 38 (38) | 36 (38) | 42 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT04583618/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04583618/SAP_001.pdf